CLINICAL TRIAL: NCT05666921
Title: Somatic Symptoms, Alexithymia and Styles of Attachment: a Cross-sectional Study
Brief Title: Alexithymia and Attachment Style in Patients With Somatic Symptoms
Status: Recruiting | Type: Observational
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Rosanna Martin, Principal Investigator, Meyer Children's Hospital IRCCS
Other Study IDs: somatic symptoms
Record Dates: First submitted 2022-01-05; First posted 2022-12-28 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Somatic Symptom Disorder
Keywords: somatic symptoms; alexithymia; attachment style; pain; reflective function
MeSH Terms: conditions — Medically Unexplained Symptoms; Affective Symptoms; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pediatric patients: The group is made up of pediatric patients, and an accompanying caregiver, belonging to the functional chronic pain clinic of Pain Therapy and Palliative Care, to the Gastroenterology and Nutrition Unit, to the Bronchopneumology Unit and Medical Pediatrics as well as to the Pediatric Psychology Unit, who present with somatic symptom disorders.
  Interventions: Other: psychological assessment
- Control group: The population of the control group, recruited through informal channels according to a sampling of convenience, will be enrolled on the basis of the expected inclusion criteria.
  Interventions: Other: psychological assessment

INTERVENTIONS:
Other: psychological assessment — The intervention consists in the assessment of some psychological aspects (emotional awareness, attachment style and the ability to abstract and symbolize (IQ)) of pediatric patients who present with somatic symptom disorders. , through specific tests. Each patient fills out the test battery during the psychological consult. At the same time, it is involved a parent to collect personal and clinical data through an ad hoc questionnaire.

SUMMARY:
To evaluate whether emotional awareness, attachment style and the ability to abstract and symbolize (IQ) influence the appearance of somatic symptoms. Hypothesis: the investigators expect the presence of somatic symptoms linked to the lower ability of emotional awareness, to lower ability to abstract and symbolize and to an insecure attachment style.

DETAILED DESCRIPTION:
Somatic Symptom Disorder (eg pain, weakness, chronic fatigue) represents one of the main reasons why patients seek specialist medical advice. Although the symptoms often manifest themselves in a disabling form and there are numerous medical examinations to which patients undergo, these do not seem to find an organic confirmation to their problem and consequently the patients do not receive a specific diagnosis. These are usually transient symptoms but it can happen that they become persistent and chronic, going to constitute themselves as real somatic syndromes. The study investigates the psychological and family aspects that seem to characterize somatic and chronic pain symptoms in pediatric age. In addition to this objective, the study aims to quantify the health costs incurred in the diagnostic phase prior to the classification of the somatic symptom. These elements would make it possible to achieve greater knowledge of clinical pictures and the identification of useful markers for the clinician to make early diagnoses and guide patients in a global and timely care.

ELIGIBILITY:
Inclusion Criteria:

* Clinical condition characterized by somatic symptoms such as recurrent abdominal pain, recurrent vomiting, dyspepsia, psychogenic cough, and chronic functional pain (headache, migraine, musculoskeletal pain) for which an organic cause has been excluded and whose symptom has had a strong impact on the quality of life (presence of the symptom for six months, school absenteeism, social isolation, immobility, psychological distress, difficulty in participating in sports and extracurricular activities, etc.), as per Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria.
* Age between 11 and 17 years
* Italian speaking
* Patients' and parents' consent

Exclusion Criteria:

* Cognitive and/or developmental impairment
* Difficulty in understanding the Italian language
* Presence of organic disease diagnosis
* Lack of informed consent
* Patient who does not meet DSM-5 criteria for somatic symptom disorder

Caregiver exclusion criteria:

* Cognitive deficits
* Difficulty in understanding the Italian language
* Lack of informed consent

Control group population inclusion criteria:

* Age between 11 and 17 years
* Adequate knowledge of the Italian language
* Consent to participate

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The population under study is made up of pediatric patients (aged from 11 to 17), and an accompanying caregiver, belonging to the functional chronic pain clinic of Pain Therapy and Palliative Care, to the SOC of Gastroenterology and Nutrition, to the SOSA of Bronchopneumology and to the SOC of Medical Pediatrics as well as to the SOSA of Pediatric Hospital Psychology who present with somatic symptom disorders. All consecutive patients and accompanying caregivers who access the aforementioned services and who meet the expected inclusion criteria will be enrolled.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Emotional awareness | Patients fill out the questionnaire at their enrollment in the study, during their first psychological consult after medical referral.
  Emotion Awareness Questionnaire - EAQ-30 (Rieffe et al., 2008; Camodeca & Rieffe, 2013) The EAQ is a self-report test aimed at measuring the emotional awareness of children and adolescents, it is composed of 6 subscales and 30 items and has a Likert scale of 3 points. High scores obtained at the different subscales indicate a high emotional awareness. The cut offs are specific for age and sex, for the interpretation of the scores reference is made to the scores obtained by the control group in the study by Camodeca et al., 2013.
attachment style | Patients fill out the questionnaire at their enrollment in the study, during their first psychological consult after medical referral.
  The Saparation Anxiety Test - SAT, Italian version adapted from Attili (2001) is a semi-projective tool aimed at measuring the attachment style of the child and adolescent, through the analysis of reactions and verbal responses to stimuli that illustrate 6 hypothetical situations of separation by parental figures. The responses are then classified into 8 categories which calculate a score that is compared with reference score ranges that correspond to 4 different attachment styles. Specifically, scores equal to or greater than 4 indicate secure attachment, scores between 3 and 1 an ambivalent insecure attachment, scores between 0 and -2 an avoidant insecure attachment, and finally scores equal to or lower than -3 are indicative of an attachment style disorganized / confused.
Ability to abstract and symbolize (IQ) | Patients fill out the questionnaire at their enrollment in the study, during their first psychological consult after medical referral.
  Raven's Standard Progressive Matrices - SPM-RA (Raven, 1982), are a test that aims to measure the general factor of fluid intelligence. the test consists of four series (A, B, C, D) of 12 items each of increasing complexity. It is an excellent test from both a psychometric and a factorial point of view. The updated report - SPM-RA (prepared by Picone, Orsini and Pezzuti) will be used as a reference for the test scoring, which allows the instrument to be used for a sample aged 6 to 18. An intelligence score above 25/36 indicates an above average intelligence level, scores between 17/36 and 25/36 are to be considered indicative of an average intelligence level, scores below 17/36 below average intelligence medium (Picone, Orsini and Pezzuti)

SECONDARY OUTCOMES:
Stressful life events | Patients fill out the questionnaire at their enrollment in the study, during their first psychological consult after medical referral.
  Codding Life Event Scales - CLES A (Coddington, 1972) (version A for individuals aged ≥ 13). The CLES is a self-report measure that helps determine how specific events have affected a child's personal growth and adjustment. Results identify areas that may require further investigation. The scales allow clinicians to easily identify actual and potential physical and mental health problems arising from psychological causalities. By measuring significant life events in terms of Life Change Units (LCUs), the CLES can provide insight into recent events that may be affecting the respondent's health. The CLES scales also take into account the different kinds of life challenges that are faced by children of different ages. There are three scales and the items included on each refer to events that children of the particular age group may have experienced. Each form produces a Life Change Unit score that is applied to Risk Evaluation cut-off guidelines.
Behavioral and emotional issues | Parents fill out the questionnaire at their enrollment in the study, during their first psychological consult after medical referral.
  The Child Behavior Checklist - CBCL / 6-18 is a self-report test aimed at parents of children aged 6 to 18, aimed at measuring, in addition to adaptive skills, eight syndromes: Anxiety / Depression, Withdrawal / Depression, Somatic complaints, Social problems, Thinking problems, Attention problems, Rule-breaking behavior, Aggressive behavior. These syndromes represent categories of problems that tend to be associated and are organized in two superordinate scales: scale of Internalization Problems and scale of Outsourcing Problems. The standard scores are scaled so that 50 is the average for age and gender, with an sd of 10 points. Higher scores indicate greater problems. Score located below the 93rd percentile are considered to be the average, scores between the 93-97th percentile are borderline and any score above the 97th percentile is within the clinical range.
stress and protection indicators | Patients fill out the questionnaire at their enrollment in the study, during their first psychological consult after medical referral.
  The Draw-a-Person-in-the-Rain Test (DAPR) is a projective test that theoretically creates a situation for projecting a symbolic image of oneself in a stressful environment (Hammer, 1958). It measures stress factors and defense ability by drawings of a person in the rain. The DAPR uses two rating scales: the first one hypothetically measures coping resources and rates various forms of protection against the rain (eg. hat, coat, shoes or boots, an umbrella, etc); the second scale hypothetically measures stress and includes features of the rain itself (eg. large raindrops, dense rain, puddles and clouds, etc.). In addition to the two scores, a Coping Balance index is derived by subtracting the number of stress indicators from the number of protective indicators. In theory, a person with more coping resources could manage higher levels of stress without being overwhelmed.
pain coping strategies | Patients fill out the questionnaire at their enrollment in the study, during their first psychological consult after medical referral.
  The Waldron/Varni Pediatric Pain Coping Inventory (PPCI) was developed to be a standardized questionnaire to assess systematically children's pain coping strategies. The PPCI was administered to 187 children and adolescents experiencing musculoskeletal pain associated with rheumatologic diseases. A principal components analysis revealed a five-factor solution for the PPCI: (1) cognitive self-instruction, (2) seek social support, (3) strive to rest and be alone, (4) cognitive refocusing, and (5) problem-solving self-efficacy. The results of this research provide initial evidence that the PPCI is a conceptually valid and internally reliable measure for assessing pediatric pain coping strategies
Demographic and health variables | Parents fill out the questionnaire at their enrollment in the study, during their first psychological consult after medical referral.
  Questionnaire addressed to the accompanying caregiver to collect demographic and disease data together with data on patient life events
Perceived pain, duration and impact on life areas | Patients fill out the questionnaire at their enrollment in the study, during their first psychological consult after medical referral.
  Visual Analogue Scale - VAS (Scott, Ansell, & Huskisson, 1977) standardized test for pain measurement in children over 7 years of age. The child is asked to indicate, on a numbered line, the point corresponding to the pain intensity they feel: the left extremity is marked with the label "no pain" and the right extremity with "the worst possible pain". The distance, expressed in centimeters, from the left end of the scale coincides with the evaluation.
Parental Reflective Functioning | Parents fill out the questionnaire at their enrollment in the study, during their first psychological consult after medical referral.
  The Parental Reflective Functioning Questionnaire (Luyten et al., 2017) consists of two versions: PRFQ and PRFQ-A.The PRFQ (valid. It Pazzagli et al., 2018) is an 18-item questionnaire for parents and children aged 3 to 11 that evaluates the parent's ability to recognize and understand the mental states that affect the child's behavior (Rutherford et al., 2013). It consists of three subscales: pre-mentalization, certainty of mental states and interest and curiosity. The PRFQ-A is the version adapted for adolescence of the PRFQ questionnaire. It consists of 18 items and is designed for parents of children aged 12 to 18.
Reflective Functioning | Patients fill out the questionnaire at their enrollment in the study, during their first psychological consult after medical referral.
  The reflective function questionnaire for youth (Fonagy et al., 2016) is a self-report questionnaire composed of 46 items on a 6-point Likert scale that allows to evaluate the reflexive capacity of adolescents aged 12 to 17 years.
Medical and psychological factors related to pregnancy, post partum and lifestyle | Parents fill out the questionnaire at their enrollment in the study, during their first psychological consult after medical referral.
  Obstetric, Pathological and Physiological Anamnesis Questionnaire and Lifestyles Questionnaire addressed to the accompanying caregiver to detect obstetric, pathological and physiological anamnesis, data relating to pregnancy, post partum, physiological acts and related pathologies, data relating to the patient's lifestyle (e.g. sleep hygiene) and the use of technological devices.

CONTACTS AND LOCATIONS:
Overall Officials: Rosanna Martin, MSc, Principal Investigator — Meyer Children's Hospital IRCCS
Locations (2):
- Italy (2):
  - Meyer Children's Hospital, Florence, Firenze
  - IRCCS Gianna Gaslini, Genova

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Afari N, Ahumada SM, Wright LJ, Mostoufi S, Golnari G, Reis V, Cuneo JG. Psychological trauma and functional somatic syndromes: a systematic review and meta-analysis. Psychosom Med. 2014 Jan;76(1):2-11. doi: 10.1097/PSY.0000000000000010. Epub 2013 Dec 12. PMID 24336429
- [Background] Andresen JM, Woolfolk RL, Allen LA, Fragoso MA, Youngerman NL, Patrick-Miller TJ, Gara MA. Physical symptoms and psychosocial correlates of somatization in pediatric primary care. Clin Pediatr (Phila). 2011 Oct;50(10):904-9. doi: 10.1177/0009922811406717. Epub 2011 May 16. PMID 21576182
- [Background] Bagby RM, Parker JD, Taylor GJ. The twenty-item Toronto Alexithymia Scale--I. Item selection and cross-validation of the factor structure. J Psychosom Res. 1994 Jan;38(1):23-32. doi: 10.1016/0022-3999(94)90005-1. PMID 8126686
- [Background] Bonvanie IJ, Kallesoe KH, Janssens KAM, Schroder A, Rosmalen JGM, Rask CU. Psychological Interventions for Children with Functional Somatic Symptoms: A Systematic Review and Meta-Analysis. J Pediatr. 2017 Aug;187:272-281.e17. doi: 10.1016/j.jpeds.2017.03.017. Epub 2017 Apr 14. PMID 28416243
- [Background] Cerutti R, Spensieri V, Valastro C, Presaghi F, Canitano R, Guidetti V. A comprehensive approach to understand somatic symptoms and their impact on emotional and psychosocial functioning in children. PLoS One. 2017 Feb 8;12(2):e0171867. doi: 10.1371/journal.pone.0171867. eCollection 2017. PMID 28178333
- [Background] Coddington RD. The significance of life events as etiologic factors in the diseases of children. II. A study of a normal population. J Psychosom Res. 1972 Jun;16(3):205-13. doi: 10.1016/0022-3999(72)90045-1. No abstract available. PMID 5072914
- [Background] Kascakova N, Furstova J, Hasto J, Madarasova Geckova A, Tavel P. The Unholy Trinity: Childhood Trauma, Adulthood Anxiety, and Long-Term Pain. Int J Environ Res Public Health. 2020 Jan 8;17(2):414. doi: 10.3390/ijerph17020414. PMID 31936285
- [Background] Friedrichsdorf SJ, Postier A, Eull D, Weidner C, Foster L, Gilbert M, Campbell F. Pain Outcomes in a US Children's Hospital: A Prospective Cross-Sectional Survey. Hosp Pediatr. 2015 Jan;5(1):18-26. doi: 10.1542/hpeds.2014-0084. PMID 25554755
- [Background] Friedrichsdorf SJ, Giordano J, Desai Dakoji K, Warmuth A, Daughtry C, Schulz CA. Chronic Pain in Children and Adolescents: Diagnosis and Treatment of Primary Pain Disorders in Head, Abdomen, Muscles and Joints. Children (Basel). 2016 Dec 10;3(4):42. doi: 10.3390/children3040042. PMID 27973405
- [Background] Fonagy P, Luyten P, Moulton-Perkins A, Lee YW, Warren F, Howard S, Ghinai R, Fearon P, Lowyck B. Development and Validation of a Self-Report Measure of Mentalizing: The Reflective Functioning Questionnaire. PLoS One. 2016 Jul 8;11(7):e0158678. doi: 10.1371/journal.pone.0158678. eCollection 2016. PMID 27392018
- [Background] Geist R, Weinstein M, Walker L, Campo JV. Medically unexplained symptoms in young people: The doctor's dilemma. Paediatr Child Health. 2008 Jul;13(6):487-91. PMID 19436430
- [Background] Ha C, Sharp C, Ensink K, Fonagy P, Cirino P. The measurement of reflective function in adolescents with and without borderline traits. J Adolesc. 2013 Dec;36(6):1215-23. doi: 10.1016/j.adolescence.2013.09.008. Epub 2013 Oct 25. PMID 24215968
- [Background] Janssens KA, Oldehinkel AJ, Rosmalen JG. Parental overprotection predicts the development of functional somatic symptoms in young adolescents. J Pediatr. 2009 Jun;154(6):918-23.e1. doi: 10.1016/j.jpeds.2008.12.023. Epub 2009 Feb 1. PMID 19181331
- [Background] Janssens KA, Rosmalen JG, Ormel J, van Oort FV, Oldehinkel AJ. Anxiety and depression are risk factors rather than consequences of functional somatic symptoms in a general population of adolescents: the TRAILS study. J Child Psychol Psychiatry. 2010 Mar;51(3):304-12. doi: 10.1111/j.1469-7610.2009.02174.x. Epub 2009 Sep 28. PMID 19788552
- [Background] King S, Chambers CT, Huguet A, MacNevin RC, McGrath PJ, Parker L, MacDonald AJ. The epidemiology of chronic pain in children and adolescents revisited: a systematic review. Pain. 2011 Dec;152(12):2729-2738. doi: 10.1016/j.pain.2011.07.016. PMID 22078064
- [Background] Kugler BB, Bloom M, Kaercher LB, Truax TV, Storch EA. Somatic symptoms in traumatized children and adolescents. Child Psychiatry Hum Dev. 2012 Oct;43(5):661-73. doi: 10.1007/s10578-012-0289-y. PMID 22395849
- [Background] Luyten P, Mayes LC, Nijssens L, Fonagy P. The parental reflective functioning questionnaire: Development and preliminary validation. PLoS One. 2017 May 4;12(5):e0176218. doi: 10.1371/journal.pone.0176218. eCollection 2017. PMID 28472162
- [Background] Moreno MA. Functional abdominal pain in children and adolescents. JAMA Pediatr. 2013 Feb;167(2):204. doi: 10.1001/jamapediatrics.2013.1665. No abstract available. PMID 23381459
- [Background] Schulte IE, Petermann F. Somatoform disorders: 30 years of debate about criteria! What about children and adolescents? J Psychosom Res. 2011 Mar;70(3):218-28. doi: 10.1016/j.jpsychores.2010.08.005. Epub 2010 Nov 4. PMID 21334492
- [Background] Taylor EM, Boyer K, Campbell FA. Pain in hospitalized children: a prospective cross-sectional survey of pain prevalence, intensity, assessment and management in a Canadian pediatric teaching hospital. Pain Res Manag. 2008 Jan-Feb;13(1):25-32. doi: 10.1155/2008/478102. PMID 18301813
- [Background] Taylor GJ, Parker JD, Bagby RM, Acklin MW. Alexithymia and somatic complaints in psychiatric out-patients. J Psychosom Res. 1992 Jul;36(5):417-24. doi: 10.1016/0022-3999(92)90002-j. PMID 1619582
- [Background] Troisi A, D'Argenio A, Peracchio F, Petti P. Insecure attachment and alexithymia in young men with mood symptoms. J Nerv Ment Dis. 2001 May;189(5):311-6. doi: 10.1097/00005053-200105000-00007. PMID 11379975
- [Background] van der Veek SM, Derkx HH, de Haan E, Benninga MA, Boer F. Emotion awareness and coping in children with functional abdominal pain: a controlled study. Soc Sci Med. 2012 Jan;74(2):112-9. doi: 10.1016/j.socscimed.2011.10.023. Epub 2011 Nov 27. PMID 22196250
- [Background] Varni JW, Waldron SA, Gragg RA, Rapoff MA, Bernstein BH, Lindsley CB, Newcomb MD. Development of the Waldron/Varni pediatric pain coping inventory. Pain. 1996 Sep;67(1):141-150. doi: 10.1016/0304-3959(96)03077-1. PMID 8895242
- [Background] Wearden AJ, Lamberton N, Crook N, Walsh V. Adult attachment, alexithymia, and symptom reporting: an extension to the four category model of attachment. J Psychosom Res. 2005 Mar;58(3):279-88. doi: 10.1016/j.jpsychores.2004.09.010. PMID 15865953